CLINICAL TRIAL: NCT05347940
Title: EFFICACY OF MIRROR THERAPY IN IMPROVING HAND FUNCTION POST FLEXOR TENDON REPAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed mohamed nagy, lecturer of physical therapy for surgery- cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003533
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Hand Tendon Injury
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: 30 adult of both sexes will participate in this study and selected from outpatient clinic of faculty of physical therapy Cairo university. Their ages range from 20 to 45 years.
  Informed consent will be taken from all patients.
  All the adult were divided into two groups of equal number (15):
  Study group (A): received traditional physical therapy program in addition to motor imagery in form of mirror therapy.
  Study group (B): received traditional physical therapy program only.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (A) (Experimental): Study group (A):15 patient received traditional physical therapy program in addition to motor imagery in form of mirror therapy.
  Interventions: Other: mirror therapy
- Study group (B) (Experimental): Study group (B):15 patient received traditional physical therapy program only.
  Interventions: Other: traditional physiotherapy protocol for flexor tendon repair

INTERVENTIONS:
Other: mirror therapy — A Mirror box will be used to easily create illusion. It' is a box with one mirror in the center where on each side of it, the hands are placed in a manner that the affected limb is kept covered always and the unaffected limb is kept on the other side whose reflection can be seen on the mirror.
  Arms: Study group (A)
Other: traditional physiotherapy protocol for flexor tendon repair — include stretching exercises and active ROM exercises
  Arms: Study group (B)

SUMMARY:
This current study will be designed to prove the therapeutic effect of mirror therapy on physical function of the hand after flexor tendon repair

DETAILED DESCRIPTION:
Purpose of the study are to clarify the effectiveness of mirror therapy (MT) on pain, range of motion and hand function in post tendons repair patients. 30 adult of both sexes will participate in this study and selected from outpatient clinic of faculty of physical therapy Cairo university. Their ages range from 20 to 45 years.

Informed consent will be taken from all patients. All the adult were divided into two groups of equal number (15) Study group (A): received traditional physical therapy program in addition to motor imagery in form of mirror therapy.

Study group (B): received traditional physical therapy program only.

Procedures of the study:

* A verbal explanation about the importance of this study procedures, main aims and conceptual approach were explained to every patient.
* The procedures of this study will be divided into two main categories:

Measurement procedures:

1. Preparatory phase

   In this phase, each patient was achieved the following steps:
   * All participants will be signed an institutional review board approved informed consent statement prior to testing.
   * Subjects will be familiarized with equipment and test procedures before testing commenced.
   * All patients will be given an explanatory session before the evaluation procedure based on the protocols set.

   Primary brief medical history had been obtained, and demographic data had been recorded, including age, sex, height, weight, general health status, and activity level to decide if the patient was able to undergo the experiment.
   * Each subject's history will be taken carefully to collect information about his general condition, physical activity and current medication.
   * Measurements will be performed under standardized conditions as the following:

   Measurements will be carried out by the same investigator.

   -The measurements procedures will be conducted two times, before treatment application (pre-treatment) and after eight weeks of treatment application (post-treatment).

   Patients will be introduced to the lab at the scheduled dates, had taken the general knowledge about the system, and revised the evaluation procedures prior to onset of evaluation.

   Each subject will be tested in a single session.
2. Measuring phase

   * Standard geniometer to measure Active ROM.
   * Michigan Hand Questionnaire for hand function.
   * Visual analog scale for pain assessment.

Therapeutic procedures:

This current study will be designed to prove the therapeutic effect of mirror therapy on physical function of the hand after flexor tendon repair, so the treatment protocol will be applied through the following steps and phases:

Therapeutic intervention for the study was started at the same time for all groups of the study as following;

Exercise therapy protocol:

1. Preparatory phase

   Preparation of the patients:

   The patients will be checked carefully to make sure there will be no contraindications.

   Every patient will be given information about the measurement and treatment procedures before the beginning of the treatment.

   All participants will be asked to be cooperating with treatment program.
2. Application phase:

Mirror therapy :

A Mirror box will be used to easily create illusion. It' is a box with one mirror in the center where on each side of it, the hands are placed in a manner that the affected limb is kept covered always and the unaffected limb is kept on the other side whose reflection can be seen on the mirror.

Mirror therapy will be performed for 30 min 3 times per week for 8 weeks

ELIGIBILITY:
Inclusion Criteria:

Age 20-45 Males and females Flexor tendons repair All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

Open fractures Associated vascular injury Cruch injuries Cognitive disorders

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-05 (Estimated); Primary Completion 2022-07-22 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Active ROM | 8 weeks
  Active ROM of the finger with repaired tendon using Standard geniometer
Hand function | 8 weeks
  Hand function using Michigan Hand Questionnaire
pain assessment | 8 weeks
  pain assessment using Visual analog scale

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University, Giza
  - Cairo university, Giza

IPD SHARING:
Plan to Share IPD: No